CLINICAL TRIAL: NCT02973659
Title: The Use of Topical Oxybutynin 10% for Treating Primary Focal Hyperhidrosis-axillary, Palmar and Plantar.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, DERMATOLOGIST, HEAD, CENTER OF AESTHETIC DERMATOLOGY, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0471-14-TLV
Record Dates: First submitted 2016-11-06; First posted 2016-11-25 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — oxybutynin; Cholinergic Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- patients with palmar hyperhidrosis (Experimental): oxybutynin Vs placebo
  Interventions: Drug: Oxybutynin; Drug: Placebos
- patients with plantar hyperhidrosis (Experimental): oxybutynin Vs placebo
  Interventions: Drug: Oxybutynin; Drug: Placebos
- patients with axillary hyperhidrosis (Experimental): oxybutynin Vs placebo
  Interventions: Drug: Oxybutynin; Drug: Placebos

INTERVENTIONS:
Drug: Oxybutynin — 10% oxybutynin gel (one side) Vs placebo aqueous gel (other side) - 2/d application, 1 month
  Other Names: anti cholinergic
Drug: Placebos

SUMMARY:
Primary focal hyperhidrosis interferes with daily activities. Limited efficacy, costs, side effects and complications are issues of concern for most current therapeutic modalities. In this study the invetigators aim to evaluate the efficacy of topical oxybutynin 10% gel in treating primary focal hyperhidrosis. 60 patients with primary focal hyperhidrosis will be recruited. Topical oxybutynin 10% gel will be assigned to the right or left axilla, palm or sole and a placebo compound to the contralateral side for a total of 30 days. The Hyperhidrosis Disease Severity Scale (HDSS) and Dermatology Life Quality Index (DLQI) questionnaires will be administered before and after treatment, and 2 noninvolved blinded physicians will score the results using starch-iodine tests. The participants will grade the sweat reduction on both sides and rated their satisfaction.

DETAILED DESCRIPTION:
This study will be performed at the Tel Aviv Medical Center. Written informed consent will be obtained from all 60 participants prior to entering the study. patients with primary focal hyperhidrosis (palmar hyperhidrosis, axillary hyperhidrosis, plantar hyperhidrosis) who receive no topical or oral anticholinergics, iontophoresis treatment or botulinum toxin injections during the 6 months prior to study entry and did not undergone sympathectomy will be recruited. Demographic data, including gender, age and medical history will be collected before enrollment in the study, and the following patients will be excluded: pregnant or lactating women, individuals with conditions that may cause secondary hyperhidrosis, individuals with a history of eczema, seborrhea, psoriasis, glaucoma, micturition disorder, gastric retention, myasthenia gravis, angioedema, Sjögren's syndrome, or Sicca syndrome, and candidates older than 60 years or younger than 18 years.

The study will follow a prospective, randomized, double blind, placebo-controlled design. Each participant will be given a pair of test jars (designated as "'gel A"' and "'gel B"'). The investigators will use a designated software to randomize the jars (either A or B) which contained 10% oxybutynin gel or a placebo aqueous gel. The two jars are identical in shape, size and weight, as well as color, odor and consistency. The patients will be instructed to apply 1 cm of gel A or B on clean, dry and intact skin of one sweating area (right or left palms, soles or axillae) twice daily for 30 days. In addition, the participants will be instructed to avoid contact of the gel with the eyes, nose, mouth, and not to wash the areas for 4 hours post-application. The participants will be also instructed not to use any concomitant topical or systemic medication during the entire treatment period. Each jar will be weighed by a digital scale before treatment initiation and on the 30th day of treatment.

The participants will interviewed twice, first at the time of screening before the initial application and then following the completion of the 30th day of treatment. The participants will be asked to rate the severity of their condition using the hyperhidrosis disease severity scale in which a score of 3 or 4 indicates severe hyperhidrosis while a score of 1 or 2 indicates mild or moderate hyperhidrosis. The therapeutic results will be considered as "excellent" or "good" if the patient indicate a reduction of 2 or 1 points, respectively, on the HDSS score.

In addition, quality of life will be assessed by a modified Dermatology Life Quality Index. The maximum score is 30, with 0 indicating a negligible effect of the disorder on the patient's quality of life and 30 indicating a significant impact. A change of 0-1 point on the mDLQI score will be interpreted as reflecting no effect on the patient's life, a change of 2-5 points as a small effect, 6-10 points as a moderate effect, 11-20 points as a very significant modification, and 21-30 points as the most significant impact possible.

At the end of the treatment, patients will complete a questionnaire evaluating the following:

1. Sweat reduction in the treated and in the control sweating areas (0 = no change, 1 = poor (limited improvement with the patient being very much aware of sweating), 2 = fair (marked improvement, with noticeable sweating under stressful conditions only, 3 = good (marked improvement with minimal sweating under stressful conditions), and 4 = excellent improvement, with cessation of sweating)
2. Global patient satisfaction (0 = dissatisfied, 1 = partially satisfied, 2 = satisfied, and 3 = highly satisfied).
3. Side effects: dry mouth, headache, dizziness, urine retention, constipation and application site reactions (pruritus or dermatitis).

All patients will undergo the Minor iodine-starch test. The tested area will be photographed under standard conditions using the Galaxy Camera (3G) EK-GC100 photography system. Photographs taken before and after 30 days of treatment will be independently assessed by two dermatologists who are unaware of the study design. All pairs of photographs will be graded as 0 = no change, 1 = minor change of <25%, 2 = moderate change between 25-50%, 3 = major change between 50-75%, and 4 = absence or near absence of sweating.

Both the study and control gels will be compounded in an Israeli compounding pharmacy.

Continuous variables will be fed into a tabular format as means ± standard errors and compared using the Wilcoxon paired test. Categorical variables will be tested using the Fisher exact test. Correlation between raters will evaluated using Spearman's correlation. All analyses were carried out using SPSS 23.0.2.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* primary hyperhidrosis (axillary, palmar, plantar) diagnosed according to the recommended criteria4 : focal, visible and excessive sweating of at least 6 months duration without apparent cause, with at least two of the following characteristics: bilateral and symmetric, impairing daily activity, more than one episode per week, onset before age of 25 years, positive family history, cessation during sleep.
* given written informed patient consent of participation in the study

Exclusion Criteria:

* known history of conditions that may cause secondary hyperhidrosis
* eczema, seborrhea, psoriasis
* any other active lesion on treatment site
* any treatment for hyperhidrosis within 4 weeks
* Any medical condition that can be aggravated by anticholinergic medications: glaucoma, micturition disorders, gastric retention, myasthenia gravis, angioedema , known history of Sjögren's syndrome or Sicca syndrome
* iodine allergy
* lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The change of Dermatology Life Quality Index (DLQI) | baseline and following 30 days
the chanhe of Hyperhidrosis Disease Severity Scale (HDSS) | baseline and following 30 days

SECONDARY OUTCOMES:
sweat reduction grading | 30 days
satisfaction rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Artzi, MD, Principal Investigator — Dermatology department Tel Aviv medical center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schollhammer M, Brenaut E, Menard-Andivot N, Pillette-Delarue M, Zagnoli A, Chassain-Le Lay M, Sassolas B, Jouan N, Le Ru Y, Abasq-Thomas C, Greco M, Penven K, Roguedas-Contios AM, Dupre-Goetghebeur D, Gouedard C, Misery L, Le Gal G. Oxybutynin as a treatment for generalized hyperhidrosis: a randomized, placebo-controlled trial. Br J Dermatol. 2015 Nov;173(5):1163-8. doi: 10.1111/bjd.13973. Epub 2015 Oct 14. PMID 26114588
- [Result] Wolosker N, de Campos JR, Kauffman P, Puech-Leao P. A randomized placebo-controlled trial of oxybutynin for the initial treatment of palmar and axillary hyperhidrosis. J Vasc Surg. 2012 Jun;55(6):1696-700. doi: 10.1016/j.jvs.2011.12.039. Epub 2012 Feb 16. PMID 22341836
- [Result] Try C, Messikh R, Elkhyat A, Aubin F, Humbert RP. [Use of oral oxybutynin at 7.5 mg per day in primary hyperhidrosis]. Rev Med Liege. 2012 Oct;67(10):520-6. French. PMID 23167161
- [Result] Cartwright R, Srikrishna S, Cardozo L, Robinson D. Patient-selected goals in overactive bladder: a placebo controlled randomized double-blind trial of transdermal oxybutynin for the treatment of urgency and urge incontinence. BJU Int. 2011 Jan;107(1):70-6. doi: 10.1111/j.1464-410X.2010.09508.x. PMID 20626389
- [Result] Sand PK, Davila GW, Lucente VR, Thomas H, Caramelli KE, Hoel G. Efficacy and safety of oxybutynin chloride topical gel for women with overactive bladder syndrome. Am J Obstet Gynecol. 2012 Feb;206(2):168.e1-6. doi: 10.1016/j.ajog.2011.08.005. Epub 2011 Aug 11. PMID 21963104
- [Result] Staskin DR, Dmochowski RR, Sand PK, Macdiarmid SA, Caramelli KE, Thomas H, Hoel G. Efficacy and safety of oxybutynin chloride topical gel for overactive bladder: a randomized, double-blind, placebo controlled, multicenter study. J Urol. 2009 Apr;181(4):1764-72. doi: 10.1016/j.juro.2008.11.125. Epub 2009 Feb 23. PMID 19233423